CLINICAL TRIAL: NCT06027112
Title: Risk Factor Association of Musculoskeletal Injuries Among University Students
Status: Recruiting | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: 41923
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Injuries
Keywords: Posture, sleep, physical activity, demographics
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male
  Interventions: Other: musculoskeletal injuries
- Female
  Interventions: Other: musculoskeletal injuries

INTERVENTIONS:
Other: musculoskeletal injuries — This research will be conducted to identify the factors that increase the risk of musculoskeletal injuries in university students,

SUMMARY:
This research will be conducted to identify the factors that increase the risk of musculoskeletal injuries in college students, Hypothesis: Demographic, anthropometric, postural, sleep quality and physical activity characteristics significantly predicted musculoskeletal injury.

DETAILED DESCRIPTION:
An important public health issues for young people, particularly university students is musculoskeletal injuries.The wound may cause excruciating agony, functional limitations,and decreased quality of life (Almeida et al.,2013). musculoskeletal injuries have a complicated etiology, with important roles played by demographics, anthropometric, psychological,postural, sleep quality, and physical activity variable.To create focused preventives and intervention measures, it is essential to understand the risk factor of musculoskeletal injuries among university students.

Questionnaire has been extensively utilized to asses postural risk factor for musculoskeletal illness such as low back pain. Musculoskeletal injuries have been linked to possible risk factors related to sleep quality, physical activity in previous study. However it is still unclear how these factor interact in a complex way and how that affects the likelihood of musculoskeletal injury.

By examining the association between demographics, anthropometric, phycological, postural, sleep quality and physical activity in university students,this study seeks to fill this vacuum in the literature.The results of this study will offer insightfull information that will help to guide the creation of focused preventives and intervention for this demographics.

The date will be collected through the use of structure questionnaire the survey will ask questions on demographics data, psychological aspects, posture, sleep patterns, and level of physical activity and the participants will be required to complete the 9-test screening Battery for musculoskeletal damage.

The following resources will be utilized to gather information on various aspects of musculoskeletal injuries.

Age, gender, height, weight, and body mass index (BMI) General health questionnaire (GHQ) Nordic musculoskeletal questionnaire for posture evaluation (NMQ) Pittsburgh sleep quality index is used to evaluate sleep quality (pSQI) International physical activity questionnaire for measuring physical activity (IPAQ) Screening for musculoskeletal injuries:9-test MSK injury screening Battery

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate students
* ages of 18 and 25.

Exclusion Criteria:

* Graduate students
* younger than 18 or older than 25
* who refuse to take part in the study will all be disqualified.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate students who are willing to engage in the study must be between the ages of 18 and 25.
Sampling Method: Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Risk Factor Association of Musculoskeletal Injuries Among University Students | 3 Months
  yes/NO

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Ict, Pakistan

IPD SHARING:
Plan to Share IPD: No